CLINICAL TRIAL: NCT02715141
Title: Molecular Stool Testing for Colorectal Cancer Surveillance
Acronym: MOCCAS
Status: Completed | Type: Observational
Sponsor: The Netherlands Cancer Institute (Other)
Collaborators: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: M15MOC; NL52708.018.15 (Other: CCMO, the Netherlands)
Record Dates: First submitted 2016-02-17; First posted 2016-03-22 (Estimated); Last update posted 2022-01-25 (Actual); Status verified 2022-01

CONDITIONS: Colorectal Cancer
Keywords: surveillance, molecular stool testing
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Stool samples will be collected. The stool samples will be used to test for the presence of molecular stool markers.
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Collection of stool sample — Collection of stool sample prior to the scheduled surveillance colonoscopy.

SUMMARY:
Rationale: Since January 2014 the Dutch screening programme for bowel cancer has been implemented. Screening will increase the demand for surveillance. Although patients in whom adenomas have been removed are at increased risk of progressing to cancer, solid evidence on the reduction of death from CRC through the current colonoscopy-based surveillance is lacking. Furthermore, colonoscopy-based surveillance leads to high logistic demands, high individual burden and high costs. Therefore, there is need for new surveillance strategies. Stool-based molecular testing (Cologuard®, consisting of a stool DNA test and an immunochemical assay for human hemoglobin) or Faecal Immunochemical Testing (FIT) may serve as an alternative for colonoscopy surveillance.

The aim of this study is to compare the accuracy of an established molecular stool test (Cologuard®) and FIT to colonoscopy for detection of advanced adenomas or CRC (advanced neoplasia) in a surveillance population. These outcomes will be used to model various strategies of stool-based molecular surveillance to inform health policy decisions.

DETAILED DESCRIPTION:
BACKGROUND: Since January 2014 the Dutch screening programme for colorectal carcinoma (CRC) has been implemented. Screening will increase the demand for surveillance. However, solid evidence on the reduction of death from CRC through the current colonoscopy-based surveillance is lacking. Furthermore, colonoscopy-based surveillance leads to high logistic demands, high patient burden and high costs. Therefore, there is need for new surveillance strategies. Stool-based molecular testing (Cologuard®) or Faecal Immunochemical Testing (FIT) may serve as an alternative for colonoscopy surveillance.

OBJECTIVES:

1. To compare the accuracy of an established molecular stool test (Cologuard®) and FIT to colonoscopy for detection of advanced adenomas or CRC (advanced neoplasia) in a surveillance population.
2. To model various strategies of stool-based molecular surveillance to inform health policy decisions.

MATERIALS AND METHODS: In this prospective observational cross-sectional cohort study, individuals aged 50-75 years that are scheduled for surveillance colonoscopy will be invited to participate. They are asked to collect a whole-stool sample prior to the surveillance colonoscopy. The sample will be used to test for the presence of molecular stool markers. The results of the molecular stool test and FIT will be compared to the colonoscopy findings.

EXPECTED RESULTS: Frequent surveillance using stool-based molecular testing is more cost-effective than the current colonoscopy-based surveillance.

ELIGIBILITY:
Inclusion Criteria:

* Subjects in the age group 50-75 years. The lower age limit is set at 50 years because of the high probability of familiar predisposition when advanced neoplasm is present in a younger age group.26 The upper age limit of 75 years is in correspondence with the recommended stop-age for surveillance according to the current guideline.9
* Subjects with an indication for surveillance colonoscopy according to the previous guideline ('Follow up after polypectomy', 2002; summarized in 2008) or current ('Colonoscopy Surveillance', 2013) guideline. This includes subjects with a history of CRC or polypectomy, as well as subjects under surveillance for familial colorectal carcinoma (FCC).
* Subjects who have sufficient comprehension of the Dutch language.
* Subjects who have given their informed consent.

Exclusion criteria:

* Subjects with inflammatory bowel disease (IBD)
* Subjects with Lynch syndrome, familial adenomatous polyposis (FAP), attenuated FAP (AFAP), MUTYH associated polyposis (MAP) and serrated polyposis syndrome (SPS)
* Subjects with a previous colonoscopy < 6 months (rescopy)
* Subjects with proctocolectomy
* Subjects with life expectancy < 3 years

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The intended population of this study consists all subjects in the participating centres that are elected for colonoscopy surveillance.
Sampling Method: Non-Probability Sample
Enrollment: 3966 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2020-12-15 (Actual)

PRIMARY OUTCOMES:
accuracy of molecular stool test (Cologuard) and FIT | Patient inclusion for the calculation of the accuracies is expected to take 2-3 years.
  The accuracy (sensitivity, specificity, PPV and NPV) of the molecular stool test (Cologuard®) and FIT compared to colonoscopy in the detection of advanced neoplasia in a surveillance population.
cost-effectiveness of stool-based surveillance strategies using the ASCCA (Adenoma and Serrated pathway to Colorectal CAncer) model | This will be calculated when all accuracy data (outcome 1) are available. This is expected to be 6 months after end of study.
  Cost-effectiveness of multiple surveillance strategies, using test performance data as input in the ASCCA (Adenoma and Serrated pathway to Colorectal CAncer) model.
life time health effects of stool-based surveillance strategies using the ASCCA (Adenoma and Serrated pathway to Colorectal CAncer) model | This will be calculated when all accuracy data (outcome 1) are available. This is expected to be 6 months after end of study.
  The ASCCA model will be used to predict outcomes, including cancer incidence and mortality, for different surveillance strategies.

SECONDARY OUTCOMES:
risk of CRC | up to one month after surveillance colonoscopy
  Risk factors for detecting advanced colonic neoplasia have been identified, of which the most established include gender, age, BMI, family history, physical activity, nutritional habits and smoking. Participants will be asked to complete a validated online questionnaire evaluating these risk factors.
presence of Cologuard marker pannel on resected tissue of polyps | Analysis will be performed during the study and approximately 1 year after end of study
  A challenge associated with the use of molecular markers is to find a panel of markers that represents the heterogeneity of the tumour. Therefore it is of interest to analyse whether the markers included in the Cologuard are present in the tissue of resected polyps.
presence of previously identified progression biomarker on resected tissue samples of polyps | Analysis will be performed during the study and approximately 1 year after end of study
  The identification of biomarkers involved in the progression from colorectal adenoma to carcinoma (progression biomarkers) could aid better risk-stratification of adenomas and thereby decrease over-diagnosis and over-treatment . As a secondary objective we will therefore analyse previously identified progression biomarkers in the tissue samples of polyps obtained during colonoscopy.

CONTACTS AND LOCATIONS:
Locations (1):
- Nethelands Cancer Institute, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Carvalho B, de Klaver W, van Wifferen F, van Lanschot MCJ, van Wetering AJP, van der Zander QEW, Lemmens M, Bolijn AS, Tijssen M, Delis-van Diemen P, Buekers N, Daenen K, van der Meer J, van Mulligen PG, Hijmans BS, de Ridder S, Meiqari L, Bierkens M, van der Hulst RWM, Kuyvenhoven JPH, van Berkel AM, Depla ACTM, van Leerdam ME, Jansen JM, Wientjes CA, Straathof JWA, Keulen ETP, Ramsoekh D, Moons LMG, Zacherl M, Masclee AAM, de Wit M, Greuter MJE, van Engeland M, Dekker E, Coupe VMH, Meijer GA. Stool-Based Testing for Post-Polypectomy Colorectal Cancer Surveillance Safely Reduces Colonoscopies: The MOCCAS Study. Gastroenterology. 2025 Jan;168(1):121-135.e16. doi: 10.1053/j.gastro.2024.08.022. Epub 2024 Aug 30. PMID 39218164
- [Derived] van Lanschot MC, Carvalho B, Coupe VM, van Engeland M, Dekker E, Meijer GA. Molecular stool testing as an alternative for surveillance colonoscopy: a cross-sectional cohort study. BMC Cancer. 2017 Feb 7;17(1):116. doi: 10.1186/s12885-017-3078-y. PMID 28173852